CLINICAL TRIAL: NCT07166991
Title: Impact of a Specific Anesthetic Strategy on Intraoperative Hemodynamic Stability During Organ Procurement in Brain Dead Donor: An Open-label Multicenter Randomized and Controlled Trial
Brief Title: Anesthesia sTrategy foR Organ Procurement In braiN dEath
Acronym: ATROPINE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38RC24.0238
Record Dates: First submitted 2025-05-21; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Brain-dead Organ Donors
Keywords: brain-dead organ donors; anesthesia; hemodynamic stability; sevoflurane; volatile anesthesia; sufentanil; opioid agents; organ procurement; organ harvesting; donor management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Volatile anesthetic group (Experimental): Sevoflurane administration during the organ procurement procedure
  Interventions: Drug: Volatile anesthetic; Other: Intraoperative brain-dead donor management
- Opioid anesthetic group (Active Comparator): Sufentanil administration during the organ procurement procedure
  Interventions: Drug: Opioid Anesthesia; Other: Intraoperative brain-dead donor management
- No anesthetic drug group (Active Comparator): No hypnotic (volatil anesthetics or intravenous anesthetics) or analgesic (opioid agents) drug administration during the organ procurement procedure
  Interventions: Other: Intraoperative brain-dead donor management

INTERVENTIONS:
Drug: Volatile anesthetic — In the volatile anesthetic group, sevoflurane will be administrated during the organ procurement procedure. Administration will be initiated progressively after moving in the operating room and will be pursued until aortic clamping (targeted end-expiratory concentration suggested between 1 and 2%).
  No opioid agent (or intravenous hypnotic agent) will be allowed in this group.
  Arms: Volatile anesthetic group
Drug: Opioid Anesthesia — In the opioid anesthetic group, intravenous sufentanil will be administrated during the organ procurement procedure. Continuous administration will be initiated after moving in the operating room (suggested dosage : 0,3 µg/kg/h) with supplemental dose if needed (at the discretion of the anesthesia team) and will be pursued until aortic clamping. No hypnotic drug administration will be allowed in this group.
  Arms: Opioid anesthetic group
Other: Intraoperative brain-dead donor management — In all groups (experimental and control groups), neuromuscular blocking agents will be administered during the entire procedure, according to national guidelines. In all groups, hemodynamic management (use of vasoactive agents as vasopressors or anti-hypertensive drugs) will be done according to the discretion of the anesthesia team.
  In all groups, all the others aspects of the donor management will be not modified by the study protocol.

SUMMARY:
The optimal anesthetic strategy during organ procurement in brain-dead donors remains unknown. The administration of anesthetic drugs in this setting aims to preserve hemodynamic stability in the face of reflex responses mediated by preserved spinal activity. Volatile anesthetics may blunt these reflexes, but their potential benefits in this context have never been investigated.

This randomized trial evaluates the effects of volatile anesthesia (sevoflurane), opioid administration (sufentanil), or no anesthetic drugs on intraoperative hemodynamic stability during organ procurement in brain-dead donors. The primary outcome is the proportion of operative time within a predefined arterial blood pressure range.

DETAILED DESCRIPTION:
Brain-dead donors (BDD) remain the primary source of grafts for organ transplantation in France and worldwide. The main objective of BDD management, from the diagnosis of brain death in the intensive care unit (ICU) to organ procurement (OP) in the operating room, is to restore or maintain physiological homeostasis in order to preserve graft viability and improve long-term recipient outcomes. ICU management of potential BDD-particularly through donor management goals-has been shown to increase both the number and the quality of transplanted organs.

In contrast, anesthetic management of BDD during OP is less standardized, although surgical manipulation may jeopardize donor homeostasis. Hemodynamic responses to surgical stimuli (e.g., incision and visceral manipulation), such as tachycardia and marked increases in arterial blood pressure, are well described and result from preserved spinal reflexes. These reflexes, and the vasoactive drugs administered to counteract them, may cause intraoperative hemodynamic instability potentially detrimental to grafts.

Opioids have been proposed to attenuate these responses, but they have proven ineffective in suppressing catecholamine release induced by nociceptive surgical stimulation. Volatile anesthetics (in addition to potential protective effects against ischemia-reperfusion injury) may more effectively blunt these reflex responses. However, their benefits during OP in BDD have not been demonstrated. In the absence of evidence, retrospective studies and surveys in the USA and France report wide heterogeneity in anesthetic strategies used during graft harvesting. Volatile anesthetics and opioids remain the most common agents despite the lack of proven benefit compared with no anesthetic use.

This randomized controlled trial is designed to evaluate whether volatile anesthetics (sevoflurane) improve intraoperative hemodynamic stability during OP in BDD, compared with either no anesthetic use or opioid (sufentanil) administration. The hypothesis is that halogenated agents, by blunting spinally mediated hemodynamic responses to surgical stimuli, will provide greater intraoperative hemodynamic stability than no anesthetic or an opioid-based strategy.

ELIGIBILITY:
Inclusion Criteria:

* Eligible adult brain-dead donor hospitalized in intensive care unit in one of the participating center:

  * Confirmed diagnosis of brain death according to French public health code.
  * Ongoing organ donation procedure managed by the local organ procurement coordination team with confirmation of the potential procurement of at least one intra-abdominal or intra-thoracic organ.
  * Transfer to the operating room for the organ procurement procedure scheduled for the next 6 hours and anesthesia team alerted.
* Information of the patient's next of kin by the investigator and absence of opposition to research confirmed by the testimony of the next of kin according to French public health code.

Exclusion Criteria:

* Age < 18 years.
* DCD (donation after circulatory death) donors.
* Ongoing extracorporeal circulation at the time of death.
* Hemodynamic instability at the screening visit defined by a noradrenalin dose > 1 µg/kg/min.
* Contraindication to the implementation of the anesthetic interventions evaluated in the trial:

  * Prior history of opioid or volatil anesthetic agents allergy.
  * Prior personal or family history of malignant hyperthermia or history of myopathy at risk of malignant hyperthermia.
* Opposition to the research expressed by the patient during his or her lifetime and documented by the next of kin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
A hierarchical endpoint of hemodynamic stability during the organ procurement procedure | Operative time
  Proportion of intraoperative time (between initial skin incision and aortic clamping) with a mean arterial blood pressure between 65 and 75 mmHg, between the volatile anesthetic group of brain-dead donors and :
  1. The no anesthetic drug group of brain-dead donors.
  2. The opioid anesthetic group of brain-dead donors.

SECONDARY OUTCOMES:
Comparaison of the hemodynamic stability during the organ procurement procedure between the no anesthetic drug group and the opioid anesthetic group of brain-dead donors | Operative time
  Proportion of intraoperative time (between initial skin incision and aortic clamping) with a mean arterial blood pressure between 65 and 75 mmHg.
Between-group comparaison of the proportion of intraoperative time spent in hypotention | Operative time
  Relative duration of intraoperative time (from initial skin incision to aortic clamping) spent with a mean arterial pressure < 60 mmHg.
Between-group comparaison of the proportion of brain-dead donors with a hemodynamic response at initial surgical incision | Operative time
  Occurrence of an increase in systolic blood pressure ≥ 20%, within 5 minutes of the initial surgical incision, compared with the mean systolic blood pressure registered in the 1 to 5 min preceding the initial surgical incision.
Between-group comparaison of the proportion of brain-dead donors with a hemodynamic response to sternotomy | Operative time
  Occurrence of an increase in systolic blood pressure ≥ 20%, in the 5 minutes following sternotomy, compared with the mean systolic blood pressure measured in the 1 to 5 min preceding sternotomy, in the subgroup of brain-death donors who underwent an intra-thoracic organ harvesting.
Between-group comparaison of the mean arterial blood pressure variability during the organ procurement procedure | Operative time
  Intraoperative variability of the mean arterial pressure measuring using the average real variability (ARV) index of mean arterial pressure.
Between-group comparaison of the mean arterial blood pressure variability during the organ procurement procedure | Operative time
  Intraoperative variability of the mean arterial pressure measuring using the intra-individual standard deviation of mean arterial pressure measurements (SD-MAP).
Between-group comparaison of the mean dose of catecholamines administered during the organ procurement procedure | Operative time
  Intraoperative mean dose (µg/kg/min or U/min) of each catecholamine administered (noradrenaline, adrenaline, dobutamine, vasopressin) and intraoperative mean norepinephrine equivalent score.
Between-group comparaison of the total intraoperative volume of vascular filling | Operative time
  Volume by type of feeling solution during the organ procurement procedure
Between-group comparaison of the total intraoperative volume of labile blood products | Operative time
  Volume of labile blood products by type during the organ procurement procedure
Between-group comparaison of the number of organs harvested and transplanted | 24 hours
  Number of solid organs (heart, lungs, liver, kidneys) harvested and effectivelly transplanted by brain-dead donors.
Between-group comparison of the rate of delayed graft function of the kidney | 7 days post-transplant
  Delayed graft function of the kidney in the recipient defined as the need for dialysis within 7 days post-transplant.
Between-group comparison of the rate of primary lung graft dysfunction | 72 hours
  Primary lung graft dysfunction in the recipient, as defined by the French Biomedicine Agency: Existence within 72 hours post-transplant of diffuse pulmonary opacities, the severity of which is graded from 1 to 3, depending on the PaO2/FiO2 ratio (< 200, 200-300, >300) or the need for extracorporeal oxygenation (grade 3).
Between-group comparison of the rate of primary heart graft dysfunction | 24 hours
  Primary heart graft dysfunction in the recipient, as defined by the French Biomedicine Agency: left ventricular ejection fraction < 30% (ultrasound), and/or need for mechanical circulatory assistance, re-transplantation or death of the recipient within 24 hours post-transplant.
Between-group comparison of the rate of primary liver graft dysfunction | 7 days post-transplant
  Primary liver graft dysfunction in the recipient, as defined by the French Biomedicine Agency: bilirubin ≥ 10mg/dL on day 7, international normalized ratio ≥ 1.6 on day 7, and alanine or aspartate aminotransferases >2000 IU/L within the first 7 days
Describe the number of donor management goals achieved in the 12 hours prior and during the organ procurement procedure | 24 hours
  Describe the number of donor management goals achieved in the 12 hours prior and during the organ procurement procedure, including the following:
  * Heart rate between 60 and 120 /min,
  * Diuresis between 1 and 1.5 mL/kg/h,
  * PaO2 / FiO2 ratio > 250 (if lung harvested),
  * Hemoglobin > 7 g/dL (10 g/dL if intrathoracic harvesting),
  * Blood glucose between 5 and 8 mmol/L,
  * Natremia < 155 mmol/L,
  * Core temperature > 35°C.

OTHER OUTCOMES:
Comparaison the 1-year graft survival | 1 year
  The aim of the TREATED (grafT suRvival aftEr Anesthesia sTrategy in brain dEath Donors) ancillary observational study will be to compare the 1-year graft survival of the solid organ transplanted (kidney, liver, heart, lungs) according to the randomization group of the brain-death donor included in the ATROPINE trial, adjusted on the main known risks factors for 1-year graft survival for each category of solid organ.
Compare the number and type of rejection episodes that occurred for each type of transplanted organ | 1 year
  The secondary objective of the TREATED ancillary trial will be to compare the number and type of rejection episodes that occurred for each category of transplant (kidney, liver, heart, lung) in the recipients (censored at 1 year) according to the randomization group of anesthetic strategy

CONTACTS AND LOCATIONS:
Overall Officials: Benoit CHAMPIGNEULLE, MD, PhD, Principal Investigator — University Hospital, Grenoble

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fitzgerald RD, Dechtyar I, Templ E, Fridrich P, Lackner FX. Cardiovascular and catecholamine response to surgery in brain-dead organ donors. Anaesthesia. 1995 May;50(5):388-92. doi: 10.1111/j.1365-2044.1995.tb05989.x. PMID 7793540
- [Background] Conci F, Procaccio F, Arosio M, Boselli L. Viscero-somatic and viscero-visceral reflexes in brain death. J Neurol Neurosurg Psychiatry. 1986 Jun;49(6):695-8. doi: 10.1136/jnnp.49.6.695. PMID 3525756
- [Background] Wetzel RC, Setzer N, Stiff JL, Rogers MC. Hemodynamic responses in brain dead organ donor patients. Anesth Analg. 1985 Feb;64(2):125-8. PMID 3882020
- [Background] Fitzgerald RD, Hieber C, Schweitzer E, Luo A, Oczenski W, Lackner FX. Intraoperative catecholamine release in brain-dead organ donors is not suppressed by administration of fentanyl. Eur J Anaesthesiol. 2003 Dec;20(12):952-6. doi: 10.1017/s0265021503001534. PMID 14690096
- [Background] Elkins LJ. Inhalational anesthesia for organ procurement: potential indications for administering inhalational anesthesia in the brain-dead organ donor. AANA J. 2010 Aug;78(4):293-9. PMID 20879630
- [Background] Souter MJ, Eidbo E, Findlay JY, Lebovitz DJ, Moguilevitch M, Neidlinger NA, Wagener G, Paramesh AS, Niemann CU, Roberts PR, Pretto EA Jr. Organ Donor Management: Part 1. Toward a Consensus to Guide Anesthesia Services During Donation After Brain Death. Semin Cardiothorac Vasc Anesth. 2018 Jun;22(2):211-222. doi: 10.1177/1089253217749053. Epub 2017 Dec 24. PMID 29276852
- [Background] Boutin C, Vachiery-Lahaye F, Alonso S, Louart G, Bouju A, Lazarovici S, Perrigault PF, Capdevila X, Jaber S, Colson P, Jonquet O, Ripart J, Lefrant JY, Muller L; pour le groupe AzuRea. [Anaesthetic management of brain-dead for organ donation: impact on delayed graft function after kidney transplantation]. Ann Fr Anesth Reanim. 2012 May;31(5):427-36. doi: 10.1016/j.annfar.2011.11.027. Epub 2012 Apr 26. French. PMID 22541983
- [Background] Perez-Protto S, Nazemian R, Matta M, Patel P, Wagner KJ, Latifi SQ, Lebovitz DJ, Reynolds JD. The effect of inhalational anaesthesia during deceased donor organ procurement on post-transplantation graft survival. Anaesth Intensive Care. 2018 Mar;46(2):178-184. doi: 10.1177/0310057X1804600206. PMID 29519220
- [Background] Lele AV, Vail EA, O'Reilly-Shah VN, DeGraw X, Domino KB, Walters AM, Fong CT, Gomez C, Naik BI, Mori M, Schonberger R, Deshpande R, Souter MJ; MPOG Perioperative Clinical Research Committee. Identifying Variation in Intraoperative Management of Brain-Dead Organ Donors and Opportunities for Improvement: A Multicenter Perioperative Outcomes Group Analysis. Anesth Analg. 2025 Jan 1;140(1):41-50. doi: 10.1213/ANE.0000000000007001. Epub 2024 Jul 25. PMID 39167559
- [Background] Lele AV, Nair BG, Fong C, Walters AM, Souter MJ. Anesthetic Management of Brain-dead Adult and Pediatric Organ Donors: The Harborview Medical Center Experience. J Neurosurg Anesthesiol. 2022 Jan 1;34(1):e34-e39. doi: 10.1097/ANA.0000000000000683. PMID 32149890
- [Background] Champigneulle B, Neuschwander A, Bronchard R, Fave G, Josserand J, Lebas B, Bastien O, Pirracchio R; SFAR research network. Intraoperative management of brain-dead organ donors by anesthesiologists during an organ procurement procedure: results from a French survey. BMC Anesthesiol. 2019 Jun 15;19(1):108. doi: 10.1186/s12871-019-0766-y. PMID 31202272